CLINICAL TRIAL: NCT06482398
Title: Efficacy and Safety of Cream Containing Sericin and Turmeric in Psoriasis Patients
Brief Title: Cream Containing Sericin and Turmeric in Psoriasis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COA 0087/2024
Record Dates: First submitted 2024-06-21; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Sericins; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sericin extract and turmeric extract cream (Experimental): Apply the sample 2 times a day for 8 weeks
  Interventions: Drug: Sericin extract and turmeric extract cream
- Triamcinolone acetonide 1% cream (Active Comparator): Apply the sample 2 times a day for 8 weeks
  Interventions: Drug: Triamcinolone acetonide 1% Cream

INTERVENTIONS:
Drug: Sericin extract and turmeric extract cream — Apply the sample 2 times a day for 8 weeks
  Arms: Sericin extract and turmeric extract cream
Drug: Triamcinolone acetonide 1% Cream — Apply the sample 2 times a day for 8 weeks
  Arms: Triamcinolone acetonide 1% cream

SUMMARY:
Psoriasis lesion is divided into two parts. Half of the lesion will apply cream containing sericin and turmeric and another will apply steroid cream (control). The samples will be apply two times a day for 8 weeks. Psoriasis area and severity index, physician global assessment, body surface area of lesion, dermatology life quality index, Itching score, adverse reaction are evaluated before, after using the samples for 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients with body surface area of psoriasis lesion less than 10, have psoriasis area and severity index less than 10 , and no lesion at face, hands,feet, and genital area
* No topical application on psoriasis lesion at least 2 weeks
* Willing to attend the study

Exclusion Criteria:

* Uncontrolled diseases
* Allergic to sericin turmeric and steroid
* Other skin diseases
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | 8 weeks
  Physician will evaluate the psoriasis lesion using Psoriasis Area and Severity Index. The score is graded 0 to 72 (low score means less severity and high score means high severity).

SECONDARY OUTCOMES:
Physician Global Assessment | 8 weeks
  Physician will evaluate the psoriasis lesion using Physician Global Assessment score (0 to 6, 0 means completely cleared, except for possible residual nonerythematous discoloration and 6 means condition worsened).
Body surface area of lesion | 8 weeks
  Physician will evaluate body surface area of psoriasis lesion in percentage. (low percentage means the lesion area decrease and high percentage means the lesion area increase).
Dermatology Life Quality Index | 8 weeks
  Patients will assess dermatology life quality score (0 to 30, 0 means high life quality and 30 means low life quality).
Itching score | 8 weeks
  Patients will assess itching score using visual analogue scale (0 to 10, 0 means low severity and 10 means high severity).